CLINICAL TRIAL: NCT03770975
Title: Comparison of Peri-implant Soft Tissue Esthetics Around Single Delayed Implant With Immediate Provisionalization Placed in The Esthetic Zone With and Without Using Subepithelial Connective Tissue Graft: A Randomized Clinical Trial
Brief Title: Comparison of Peri Implant Soft Tissue Esthetics With Immediate Temporization With and Without Subepithelial Connective Tissue Graft
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Osama Abdelwahab Megahed, Resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dinaosamaperio
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Immediate Temporization and Soft Tissue Augmentation Around Delayed Implants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed implant placement with immediate provisionalization (Active Comparator): Single delayed implant placement in the esthetic zone with placing an immediate temporary crown placed within 48 hours after the surgery
  Interventions: Procedure: delayed implant with immediate provisionaliztion and soft tissue graft
- Implant with immediate temporization and soft tissue graft (Experimental): Single delayed implant placement in the esthetic zone with placing a subepithelial connective tissue graft buccal to the implant and immediate temporary crown within 48 hours after the surgery
  Interventions: Procedure: delayed implant placement with immediate provisionalization

INTERVENTIONS:
Procedure: delayed implant with immediate provisionaliztion and soft tissue graft — delayed implant placement in the esthetic zone with immediate provisinalization and placement of a connective tissue graft buccal
  Arms: Delayed implant placement with immediate provisionalization
Procedure: delayed implant placement with immediate provisionalization — delayed implant placement with immediate provisionalization
  Arms: Implant with immediate temporization and soft tissue graft

SUMMARY:
The aim of this study is to clinically evaluate peri-implant soft tissue esthetics around single delayed implants in the esthetic zone.

DETAILED DESCRIPTION:
To compare the efficacy of soft tissue augmentation on the peri-implant soft tissue esthetics along with immediate temporization to immediate temporization only.

Population (P): patients with a single missing tooth in the esthetic zone Intervention (I): Delayed implant placement with immediate temporization and subepithelial connective tissue graft Comparator (C): Delayed implant placement with immediate temporization Primary outcome: Pink esthetic score (PES) Time frame: 6 months Study design: Randomized controlled clinical trial

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Good medical and psychological health
3. Absence of untreated caries lesions and untreated/uncontrolled periodontal disease. If patients required periodontal treatment (non-surgical and/or surgical), this was arranged outside the study protocol and completed at least 30 days prior to the enrolment
4. Need of a single-tooth replacement in the aesthetic (incisor, canine or premolar) region
5. Willingness to sign the informed consent form

Exclusion Criteria:

1. Any known disease (not including controlled diabetes mellitus), infections or recent surgical procedures within 30 days of study initiation;
2. Chronic treatment (i.e., 2 weeks or more) with any medication known to affect oral status (e.g., phenytoin, dihydropyridine, calcium antagonists and cyclosporine) within 1 month before baseline visit;
3. Anticoagulant therapy with warfarin, clopidogrel, ticlopidine or once daily aspirin (more than 81 mg);
4. HIV or Hepatitis;
5. Physical handicaps that would interfere with the ability to perform adequate oral hygiene;
6. Alcoholism or chronic drug abuse;
7. Heavy smokers (>10/cigarettes per day);
8. Lack of adequate primary stability at implant insertion that enables immediate provisionalization (insertion torque ca 30 Ncm).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Pink Esthetic Score | 3 months post definitive prosthesis
  Pink esthetic score evaluates the soft tissue esthetics around implant supported crowns. Using a 0-1-2 scoring system, 0 being the lowest, 2 being the highest value. The maximum achievable PES is 14. 7 variables are measured: mesial and distal papillae being 0 if absent, 1 if incomplete and 2 if complete. Alveolar process, soft tissue level, contour, texture and color being 0 if major discrepancy, 1 if minor discrepancy and 2 if matches the contralateral

SECONDARY OUTCOMES:
Patient satisfaction by Visual analogue scale (VAS) | 3 months post definitive
  Patient satisfaction will be evaluated using a questionnaire which is based on a visual analog scale (VAS). A horizontal VAS bar, 100 mm long, with the right anchor labeled "much less than natural teeth" which is marked by zero and the left anchor labeled "much more" which is marked by 10 will be used. Five questions will be formulated to record the patients' satisfaction in terms of functionality and from an esthetic point of view. Participants will look in a mirror and also be viewed a photograph before recording their answers on the horizontal calibrated line.
Buccal peri-implant soft tissue thickness | 3 months post definitive
  the soft tissue thickness buccal to the implant by using an anesthesia needle and digital caliper
Recession of the buccal peri-implant mucosa | 3 months post definitive
  measured at the apical zenith of the mucosal margin on the implants after digital superimposition of the optically scanned models as the vertical distance change between the former and the new position of soft tissue margins.

CONTACTS AND LOCATIONS:
Overall Officials: Azza Ezz AlArab, PHD, Study Chair — Professor in the department of Oral Medicine and Periodontology
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdelwahab D, Ezz AlArab A, El Nahass H. Soft tissue esthetics around immediately provisionalized delayed implants with and without connective tissue graft: A randomized clinical trial pilot study. Clin Implant Dent Relat Res. 2023 Feb;25(1):11-22. doi: 10.1111/cid.13168. Epub 2022 Dec 29. PMID 36579756